CLINICAL TRIAL: NCT01739621
Title: A Phase 2, Multi-Center, Extension Study to Evaluate the Safety, Pharmacokinetics and Efficacy of Proellex® (Telapristone Acetate) Administered Vaginally in the Treatment of Premenopausal Women With Uterine Fibroids Who Have Completed ZPV-200
Brief Title: Safety, Pharmacokinetics and Efficacy of Proellex® (Telapristone Acetate) Administered Vaginally in the Treatment of Premenopausal Women With Uterine Fibroids Who Have Completed ZPV-200
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZPV-200EXT
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Uterine Fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Proellex 12 mg (Experimental): Telapristone acetate, 1 vaginally inserted capsule, once a day, for 4 months
  Interventions: Drug: Proellex 12 mg
- Proellex 24 mg (Experimental): Telapristone acetate, 1 vaginally inserted capsule, twice a day, for 4 months
  Interventions: Drug: Proellex 24 mg

INTERVENTIONS:
Drug: Proellex 12 mg
  Other Names: telapristone acetate
  Arms: Proellex 12 mg
Drug: Proellex 24 mg
  Other Names: telapristone acetate
  Arms: Proellex 24 mg

SUMMARY:
To further determine the safety and efficacy of Proellex in premenopausal women with uterine fibroids who have previously completed study ZPV-200.

DETAILED DESCRIPTION:
This is an open label, extension study of ZPV-200 applicable to multiple study sites. Subjects will chose to administer 12 mg Proellex vaginal doses once or twice daily (morning and evening). Total study participation for ZPV-200 EXT may be up to 120 days of drug treatment separated from ZPV-200 by an off-drug interval and a 30 day follow up visit.

Subjects already enrolled in ZPV-200EXT and the remainder of the subjects who enroll will have the option of administering 12 mg vaginal capsules once or twice daily. This choice will be provided to new subjects at Visit 1.

The first 4 subjects who chose to administer 12 mg Proellex twice daily, will have additional study procedures during the baseline visit and the day after.

Once a subject has selected a dosing regimen the subject must remain on that dose for the remainder of the study.

All subjects entering the ZPV-200EXT study will have completed the ZPV-200 study and will complete an off-drug interval prior to the start of their first dosing cycle. In the off-drug interval, subject must have a menses prior to resumption of the dosing cycle in the luteal phase.

Efficacy measurements will consist of UFS-QOL (uterine fibroid symptom quality of life survey) sub-scores and total score, and number of bleeding days per drug treatment cycle as recorded in subject diaries. Fibroid size will be assessed by MRI (magnetic resonance imaging) at the end of treatment (Visit 5), and changes in size of uterine fibroids will be compared to MRI results from Visit 2 and Visit 10 of ZPV-200.

Safety measurements for this study will include adverse events (AEs), clinical laboratory tests, hormone tests, physical examinations (including breast examination and pelvic examination with PAP smear) and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Have a negative pregnancy test at the Baseline visit
* Subject has successfully completed ZPV-200 and demonstrated a return of menses

Exclusion Criteria:

* Women with abnormally high liver enzymes or liver disease. Alanine aminotransferase(ALT) or aspartate aminotransferase (AST) exceeding 1.5x upper limit normal (ULN AND)total bilirubin exceeding 1.5x ULN at baseline and confirmed on repeat).
* Clinically significant abnormal findings on baseline examination or any condition which in the opinion of the investigator would interfere with the participant's ability to comply with the study instructions or endanger the participant if she took part in the study

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Bleeding Days | 4 months
  Number of days of recorded vaginal bleeding and bleeding intensity
UFS-QOL | 4 months
  Improvements in quality of life assessed using the UFS-QOL

REFERENCES:
- See also: Corporate website — http://reprosrx.com